CLINICAL TRIAL: NCT02701504
Title: Association Between Sleep Apnea and Occurrence of Major Adverse Cardiovascular Events After Coronary Artery Bypass Grafting
Brief Title: Undiagnosed Sleep Apnea and Bypass OperaTion
Acronym: SABOT
Status: Completed | Type: Observational
Sponsor: National University of Singapore (Other)
Responsible Party: Principal Investigator, Chi-Hang Lee, Associate Professor, National University of Singapore
Other Study IDs: SABOT Study
Record Dates: First submitted 2014-09-23; First posted 2016-03-08 (Estimated); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Sleep Apnea
Keywords: sleep apnea; coronary artery bypass grafting; outcomes
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sleep apnea group: The patients who are found to have sleep apnea based on the results of the portable sleep study
- Non sleep apnea group: The patients who are found to have no sleep apnea based on the results of the portable sleep study

SUMMARY:
Sleep apnea is a prevalent disorder in patients with coronary artery disease. Previous studies suggested sleep apnea was associated with coronary plaque burden and future adverse cardiovascular events after percutaneous coronary intervention. In the SABOT study, the investigators used a FDA-approved portable sleep device to diagnose sleep apnea, and evaluate the relationship between sleep apnea and cardiovascular outcomes after non-urgent coronary artery bypass surgery.

DETAILED DESCRIPTION:
The SABOT Study is an observational study designed to study the impact of sleep apnea on cardiovascular outcomes after non-urgent coronary artery bypass surgery (CABG). Patients between the ages of 18 and 90 who are scheduled undergo an non-urgent CABG were eligible for the study

The recruited patients participants were scheduled to undergo a hospital-based overnight sleep study using a US Food and Drug Administration-approved portable monitoring devices: the Watch-PAT (Itamar Medical, Caesarea, Israel). Watch-PAT is a four-channel unattended sleep monitoring device that measures peripheral arterial tone (PAT), pulse oximetry, heart rate, and actigraphy from a built-in actigraph. Respiratory events are identified by digital vasoconstriction mediated by α-adrenergic receptors that are sensitive to surges in sympathetic activity. Respiratory events are considered to be present when one of the following three criteria was met: a reduction in PAT amplitude with an acceleration of the pulse rate or an increase in wrist activity; a reduction in PAT amplitude with ≥3% oxyhemoglobin desaturation; and ≥4% oxyhemoglobin desaturation only. Although manual scoring and editing of the Watch-PAT signals are possible, we adopted results generated by the device algorithm alone with no intervention by the operator. The diagnosis of sleep apnea is confirmed if the AHI was greater than 15 events/h.

End Points The pre-specified primary end point is a major adverse cardiac and cerebrovascular event (MACCE), defined as a composite of cardiovascular mortality, non-fatal myocardial infarction, non-fatal stroke, and repeat revascularization.

The secondary end point comprised sudden cardiac death or resuscitated cardiac arrest, all-cause mortality, and hospitalization for heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Patients with coronary artery disease scheduled to undergo non-urgent coronary artery bypass surgery

Exclusion Criteria:

* Known sleep apnea on CPAP therapy
* Cardiogenic shock on mechanical hemodynamic support
* Intubated on mechanical ventilation
* Heart failure on oxygen therapy
* Long -term alpha blocker therapy
* Severe chronic pulmonary disease
* Recurrent malignant arrhythmia
* Inability to provide informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with coronary artery disease scheduled to undergo coronary artery bypass surgery
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2013-10-01 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Major Adverse Cardiac and Cerebrovascular Events | Average of 2 years after CABG
  The number of patients with cardiac mortality, stroke, myocardial infarction, or repeat revascularization

SECONDARY OUTCOMES:
Other Cardiac and Cerebrovascular Events | Average of 2 years after CABG
  Sudden cardiac death or resuscitated cardiac arrest, all-cause mortality, hospitalization for heart failure,

CONTACTS AND LOCATIONS:
Overall Officials: Chi-Hang Lee, MD, Study Chair — National University of Singapore
Locations (1):
- National University Heart Centre, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Teo YH, Yong CL, Ou YH, Tam WW, Teo YN, Koo CY, Kojodjojo P, Lee CH. Obstructive sleep apnea and temporal changes in cardiac repolarization in patients undergoing coronary artery bypass grafting. J Clin Sleep Med. 2024 Jan 1;20(1):49-55. doi: 10.5664/jcsm.10786. PMID 38163943
- [Derived] Aung AT, Koo CY, Tam WW, Chen Z, Kristanto W, Sim HW, Kojodjojo P, Kofidis T, Lee CH. Sleep apnea and diabetes mellitus are independently associated with cardiovascular events and hospitalization for heart failure after coronary artery bypass grafting. Sci Rep. 2020 Dec 10;10(1):21664. doi: 10.1038/s41598-020-78700-9. PMID 33303900
- [Derived] Koo CY, Aung AT, Chen Z, Kristanto W, Sim HW, Tam WW, Gochuico CF, Tan KA, Kang GS, Sorokin V, Ong PJL, Kojodjojo P, Richards AM, Tan HC, Kofidis T, Lee CH. Sleep apnoea and cardiovascular outcomes after coronary artery bypass grafting. Heart. 2020 Oct;106(19):1495-1502. doi: 10.1136/heartjnl-2019-316118. Epub 2020 May 18. PMID 32423904